CLINICAL TRIAL: NCT03801785
Title: Examining the Efficacy of Pacifiers (Dummies) and Non-Nutritive Sucking (NNS) Habits in Improving Balance and Gait in 12-42 Month-Old Healthy Children Followed for 36 Months
Brief Title: Efficacy of Non-Nutritive Sucking (NNS) on Balance and Gait Measured in 12-42 Month-Old Healthy Children Over 36 Months
Acronym: NNSbenefits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Collaborators: Artsana S.p.a. (Industry)
Responsible Party: Principal Investigator, Paola Rosati, Principal Investigator (PI), Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OBG201803X004533
Record Dates: First submitted 2019-01-04; First posted 2019-01-14 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Postural Balance; Gait; Non-nutritive Sucking; Sleep; Muscle Relaxation; Electroencephalography
Keywords: Proprioceptive and exteroceptive development; Non-nutritive habit benefits; Thumb sucking; Pacifiers; Appropriate age to stop non-nutritive sucking; Dental problems; Theta Rhythm
MeSH Terms: conditions — Fingersucking | interventions — Pacifiers

STUDY DESIGN:
Intervention Model Description: The RCT includes two parallel arms. In the intervention arm, children will suck a pacifier of identical shape and type. In the control arm, children will be induced by the DDSs to stop sucking. Children's parents will be also advised by an ad hoc information sheet how to stop their children's NNS habit. Children in both arms will undergo computerized postural balancing and gait control measures every 6 months up to 36 months by video-recordings done at home or at the OBG site in Palidoro (Rome). Children in the two arms will also undergo an EEG while sucking, at enrolment and when follow-up ends. Parents will report in a diary time spent by their children on pacifier or finger-thumb sucking, crying time, afternoon and night-time sleep induction, awakenings, and day-sleep hours. Every 6 months, parents will bring the children and the diaries to the hospital. DDSs will visit the child, record oral examinations, and also report findings from parents' diaries in electronic and paper CRF.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children induced to suck pacifiers. (Experimental): Children will suck a pacifier of identical shape and type and will be allowed other NNS habits.
  Interventions: Other: Pacifier
- Children induced to stop sucking. (No Intervention): Children will be induced by DDSs to stop sucking and their parents will be advised how to stop their children's NNS habits.

INTERVENTIONS:
Other: Pacifier — The pacifiers used in this clinical trial have the same shape and material. They are produced by Artsana S.P.A. for soothing children. As such, the FDA has no jurisdictions over pacifiers (US FDA regulations May 15, 2012 https://www.fdaimports.com/blog/pacifiers-fda-change-abi-system/) because they are not medical devices intended for teething.
  Arms: Children induced to suck pacifiers.

SUMMARY:
No one disputes that fetal sucking in the womb is a natural human right. Available information on whether, how and when to stop children's sucking habits comes from popular cultural misunderstandings and lack of sound evidence-based results. Because Western countries regard thumb or pacifier (dummy) sucking after a given age as a shameful habit, parents feel stressed, anxious and even guilty for being unable to induce their children to stop non-nutritive sucking (NNS) habits or drag their unwilling child off the soothing-devices, such as pacifiers. Pacifier sucking substantially decreases the incidence of sudden infant death syndrome, reduces pain and crying, and prolongs sleeping time. Of major interest is the hypothesis that NNS improves proprioceptive and exteroceptive development including gait in big mammals (rhesus monkeys). Despite these benefits, available information claims the possible risks induced by prolonging NNS, including psychological shortfall, delayed language skills or dental problems. Despite these claims, authoritative clinical organizations worldwide reach no consensus on the appropriate age at which NNS habits should be stopped. Prompted by conflicting information from primary studies and reviews designed to balance the benefits and risks of NNS habits, our aim in this pilot open randomized controlled trial (RCT) is to test the efficacy of NNS in improving balance and gait in children enrolled at 12-42 months and followed for three years.

DETAILED DESCRIPTION:
This open pilot RCT will enroll healthy children aged 12 to 42 months coming to the Odonto-stomatology Unit at Bambino Gesù Children's Hospital and Research Institute (OBG) with their parents, who seek help in stopping their children continue the NNS habit. This RCT will last 3 years. In the first year, patient enrollment will be completed, and the analyses needed to measure the primary and secondary outcomes conducted. The RCT will test the efficacy of NNS in improving balance and gait after a two-year follow-up. Patient registries will follow internal ad hoc OBG procedures for good-clinical practice (GCP) in trial conduction (Prot. 01.01.99 published in the OBG intranet site on 5th April 2017) including patients' data registered in case report forms (CRF) in electronic and paper records. After children's parents give their consent signing the information sheet approved by the OBG Institutional Review Board (OBG-IRB), namely Comitato Etico, every eligible child will be coded with a computerized randomization code and identified in the CRF with this code, their name, surname and date of birth (RCT protocol approved on 10th September 2018, OBG-IRB Prot. N. 960). The RCT includes two parallel arms, the intervention arm and the control arm. Children in the intervention arm will suck a pacifier of identical shape and type produced by Artsana S.P.A., and will be allowed other NNS habits (finger-thumb). Children in the control arm will be induced by the OBG odonto-stomatologists (DDSs) to stop sucking and their parents will receive from the DDSs an ad hoc information sheet advising them how to stop their children's NNS habit. Children in both arms will undergo a computerized photometric postural balancing measure and gait control assessment, done by a physiotherapist (PT) delegated by the PI, every 6 months over 24 months at the Neuro-rehabilitation Unit in the OBG site at Palidoro (Rome). After enrollment, children in both arms will also undergo an electroencephalogram (EEG) while sucking, done by an EEG technician (EEG tech) delegated by the PI. Two years later, children will undergo a second EEG. Parents will report in a diary their children's time spent on pacifier or finger-thumb sucking, crying time, afternoon- and night-time sleep induction, awakenings, and daily sleeping time duration. Every 6 months, parents will bring their children and diaries to the DDSs. DDSs will visit the child and report data from oral examination findings and from parents' diaries in hospital electronic medical records and paper CRF. In accordance with the European Medicine Agency (EMA), Committee for Medicinal Products for Human Use (CHMP), International Conference on Harmonization (ICH) guidelines for GCP(EMA/CHMP/ICH/135/1995), Italian Ministry of Health law (15th July 1997) and the OBG-IRB approved RCT protocol, the OBG (acting as the Promoter for this clinical trial) and the PI are responsible for the quality assurance plan including all the enrolled children's data validation and patient registry. The PT, DDSs and the EEG tech will record also the results in an ad hoc sheet. All the variables included in the PT evaluation, orthognathic findings, parents' diary and EEGs will be recorded in an Excel file by the PT, DDSs and the EEG tech delegated by the PI. The PI is responsible for comparing and validating the data recorded and the data registered in an Excel file for the statistical analysis.

The postural balance and gait assessment, oral diagnostic examinations and EEG results detailed in every electronic and paper CRF for the children enrolled will be reviewed without undue delay by the research team including the PI, DDS members, a PT and an EEG tech delegated by the PI. These personnel will check concordance between the results and source data (electronic medical records). The PI will check, sign and date the signature on the paper CRF. If the results concern the patient's safety, the research team will inform the PI. In accordance with the OBG hospital's internal GCP protocol (Prot. OBG 01.01.11), the PI will notify adverse events to the Health Management Board and OBG-IRB. The research team will be responsible for creating a data dictionary that contains detailed descriptions of each variable used in the RCT study and CRF, including the source of the variable, coding information used and relevant ranges for outcome measures. Following the standard operating GCP procedures approved by the OBG promoter (Prot. OBG 01.01.11 and 01.01.99), the PI will archive all the documents including authorizations, contracts and all the essential documents in a trial master file in electronic and paper versions. The PI and delegate collaborators will be responsible for maintaining the CRF trace in electronic and paper forms as a locked archive in the Epidemiology Unit where the PI works. According to the internal OBG GCP procedures and always in the presence of the PI, the OBG-IRB will monitor the CRF and all documentation archived with independent monitoring activities on-site, so as to survey and assess periodically this RCT protocol and study conduction. These on-site audits will ensure that all activities related to the RCT protocol and all other data will be registered, analyzed and accurately maintained in accordance with the OBG GCP standard operating procedures specified in the foregoing. The PI will also record in the CRF every change in trial management and update the protocol in the clinicaltrial.gov website. As requested by the Italian Drug Agency, Agenzia Italiana Farmaco (AIFA), the European Medical Agency (EMA) and Food and Drug Administration (FDA), all procedures and their documentation referred to in this protocol will be made available to inspection. As specified in the aforementioned OBG GCP protocols, the electronic and paper investigator file including all the trial documentations will be kept for at least 15 years.

Sample size - Given the lack of studies investigating NNS efficacy for the primary outcome (evaluating the proprioceptive and exteroceptive benefits of NNS), to define the sample size, we analyzed the data for the incidence of instinctive NNS from all the children brought by their parents to the Odonto-stomatology Unit at Bambino Gesù Children's Hospital to investigate prolonged NNS during the year 2015. The power analysis, based on these data, estimated that 4000 children in the 12 to 42 months age group will yield an incidence rate of 2% of children (n = 80) who come for their first dental visit because of prolonged NNS. Estimating that gait (width, frequency and speed of steps, cadence, step/stride length, step/stance time, and number of falls during walking along a walkway that records spatio-temporal features) will improve in 30% of the children in the interventional arm and no children in the control arm, a study sample of 50 children will be needed to obtain a significant X2 test with α 0.05 and β of about 0.20. Assuming that 15% of the children enrolled will be lost to follow-up, sample size calculations estimate that the study needs to enroll 64 children (32 in each arm) to demonstrate a significant effect. Every 6 months after enrollment, the 64 children will attend for their dental visits. At one year after enrollment, it is estimated that reduced overbite and increased overjet, with or without stopping NNS habits, will be detected in 60 to 70% of children. It is also estimated that overbite, if present, will diminish every year by 3 mm in 40-56% of these children aged from 42 to 66 months, yielding an α of about 0.05 and β of about 0.20.

Data on outcome measures will be inserted in the RCT database progressively. Retrospective data for variables reported in the parents' diaries, or electronic and paper CRF will also be inserted in the RCT database. Missing data (unavailable, un-reported, uninterpretable or considered missing owing to data inconsistency or out-of-range results) in the RCT database will be retrieved whenever possible by the PI by interviewing parents or by re-evaluating outcome measures with PTs, DDSs or the EEG tech, and will be registered in electronic and paper CRF. Data remaining unavailable will be considered as missing.

Intellectual property and publications - Artsana S.P.A. and OBG (Promoter) signed a funding agreement (7 August 2018). They agreed that OBG is the sole owner of data and of direct and indirect RCT results. The PI is the only person responsible for the data entry and documentation archive and will follow the study as specified in the OBG-IRB protocol and its possible amendments, without disclosing any data analyses or results to Artsana S.P.A. before their publication. In future published papers, Artsana S.P.A. and OBG have agreed to state that "Artsana S.P.A. has helped to fund the RCT activities".

Practical implications and future developments - The findings obtained in this open pilot RCT should provide information on the proprioceptive, exteroceptive and muscle-relaxation benefits of NNS in children enrolled at 12 to 42 months of age and followed for 3 years (maximum age when the 3-year follow-up ends, 66 months = 5 years and 6 months). In all children follow-up will end before mixed dentition erupts.The information obtained from the EEG results should help in designing the following new research projects. For example, it will help in studies designed to identify and assess in children who prolong NNS, the pediatric population older than 36 months to enroll in a later study on diagnostic accuracy using functional magnetic resonance imaging (fMRI) without sedation (during NNS lasting at least 10 minutes) to define which neuroreceptor transmitters stimulate NNS. The fMRI findings should also help in developing a differentiated genomic analysis for girls and boys.

Statistical analysis plan - The statistical analysis will start by analyzing descriptive data for all the quantitative variables (means, medians and standard deviations) and for categorical data obtained from the electronic medical records and parents' diaries. Data frequencies and percentages will be calculated with STATA® 13 software. Various multivariate regression analyses will calculate the risk of malocclusion (Cox regression) considering as independent variables age at enrollment, sex, age at standing without support, postural balance, gait assessment and stratifying the RCT population according to possible malocclusion. The statistical significance of possible NNS-related changes in the initial malocclusion (reduced overbite and increased overjet) will be evaluated in children in whom NNS correlates with dental problems at 12, 24 and 36 months after enrollment. The statistical analysis will also assess the various types of malocclusions and correlation coefficients (r) for the psycho-social variables, including times for inducing and maintaining sleep and other variables collected in the database during a 48- to 66-month follow-up for the primary and secondary outcomes.

ELIGIBILITY:
Inclusion criteria

• Healthy boys and girls ranging in age from 12 to 42 months who tended to prolong NNS.

Exclusion criteria

* Children with craniofacial malformations or with a known or clinically suspected genetic syndrome (for example Down syndrome);
* Children with atypical swallowing for example tongue interposition, or dysphagia during swallowing caused by tongue interposition;
* Children who already have mixed dentition.

Ages: 12 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-11-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Children's postural balance force plates measured in millimeters. | Changes in postural balance assessed from date of enrollment up to 36-months.
  Multiple oscillation postural balance (swaying) measured by assessing the children's center of pressure on a stabilometric platform produced by Advanced Mechanical Technology Inc (AMTI). The X and Y axes oscillations will be aggregated by a Nexus software version 2.6 to arrive at one reported value for balance force plates in millimeters according to validated posture stability standards (Guffey et al., 2016).
Children's dynamic gait frequency assessed in steps/6-minute walking test. | Changes in gait frequency assessed from date of enrollment up to 36-months.
  Gait analysis frequency assessing children's dynamic gait steps from video recorded films. The step frequency for dynamic gait will be measured by chronometer in steps during a 6-minute walking test.
Children's step speed measured in meters/6-minute walking test. | Changes in step speed assessed from date of enrollment up to 36-months.
  Children's step speed assessed from video-recorded films during walking. The step speed will be measured by chronometer in meters during a 6-minute walking test.
Children's falls assessed as number of falls/6-minute walking test. | Changes in number of falls assessed from date of enrollment up to 36-months.
  Children's falls assessed from video-recorded films as number of falls during a 6-minute walking test.
  All the computerized photometric balance measures and gait analyses will be assessed at the Neuro-rehabilitation Unit in the OBG site at Palidoro with the PI supervision. Postural balance and gait measures will be assessed and compared with the average age-related standards.

SECONDARY OUTCOMES:
Overbite measured in millimeters during standard orthodontic assessment. | Changes in overbite from date of enrollment up to 36 months.
  DDSs will evaluate the overbite millimetric measurement calibrated for each patient and documented by intraoral photographs obtained at enrollment and every 6 months in all the children enrolled.
Overjet measured in millimeters during standard orthodontic assessment. | Changes in overjet from date of enrollment up to 36 months.
  DDSs will evaluate the overjet millimetric measurement calibrated for each patient and documented by intraoral photographs obtained at enrollment and every 6 months in all the children enrolled.
Brain areas elicitated by the NNS habit (theta-bands indicating pleasure and well-being including right and left cervico-parietal and temporo-occipital areas when children are falling asleep and sleep) recorded by EEGs at enrollment and 2 years later. | At enrollment and 2 years later.
  The EEG recorded during sucking with a pacifier or with a finger, done at enrollment and 2 years later, will identify the brain areas stimulated by NNS. These brain areas will be compared and correlated with muscle relaxation and sleep induction in the two population arms.
Awake pacifier sucking or NNS time measured in hours. | Changes in awake pacifier sucking or NNS measured from date of enrollment up to 36 months.
  Time in hours spent on awake pacifier sucking or NNS habits assessed from parents' questionnaires collected by the DDS every 6 months.
Crying time measured in minutes of crying/day. | Changes in crying time measured from date of enrollment up to 36 months.
  Time in minutes spent on crying during the day assessed from parents' questionnaires collected by the DDS every 6 months.
Sleep induction time measured in minutes/afternoon or /night-time sleep. | Changes in sleep induction measured from date of enrollment up to 36 months.
  Minutes spent on sleep induction assessed from parents' questionnaires collected by the DDS every 6 months.
Awakenings measured in number of awakenings/afternoon or /night-time sleep. | Changes in number of awakenings measured from date of enrollment up to 36 months.
  Number of awakenings during afternoon or night-time sleep assessed from parents' questionnaires collected by the DDS every 6 months.
Afternoon and night-time sleep duration measured in hours/day. | Changes in duration of afternoon or night-time sleep assessed from enrollment up to 36 months.
  Duration in hours of continuous afternoon or night-time sleep assessed from parents' questionnaires collected by the DDS every 6 months.

OTHER OUTCOMES:
Child's age in months when parents first tried to stop NNS. | At enrollment.
  Child's age in months when parents first tried to stop NNS, collected from parents by DDSs during the clinical history.
Parents' reasons for inducing children to stop NNS habits reported in a list including percentages. | At enrollment.
  Qualitative information collected from parents by DDSs during the clinical history.
How parents tried to stop NNS habits reported in a list including percentages. | At enrollment.
  Qualitative information collected from parents by DDSs during the clinical history.

CONTACTS AND LOCATIONS:
Overall Officials: Paola ROSATI, MD MSc, Principal Investigator — Bambino Gesù Children's Hospital IRCCS Rome
Locations (1):
- Bambino Gesù Children's Hospital and Research Institute, Roma, Italy

IPD SHARING:
Plan to Share IPD: No
For privacy reasons, the individual patient data (IPD) will be not shared with other researchers. At RCT completion, the PI and investigators will disseminate the statistically analyzed IPD in peer reviewed medical journals.

REFERENCES:
- [Background] Guffey K, Regier M, Mancinelli C, Pergami P. Gait parameters associated with balance in healthy 2- to 4-year-old children. Gait Posture. 2016 Jan;43:165-9. doi: 10.1016/j.gaitpost.2015.09.017. Epub 2015 Sep 30. PMID 26439183
- [Background] Lehtonen J, Valkonen-Korhonen M, Georgiadis S, Tarvainen MP, Lappi H, Niskanen JP, Paakkonen A, Karjalainen PA. Nutritive sucking induces age-specific EEG-changes in 0-24 week-old infants. Infant Behav Dev. 2016 Nov;45(Pt A):98-108. doi: 10.1016/j.infbeh.2016.10.005. Epub 2016 Oct 26. PMID 27792918
- [Background] Maulsby RL. An illustration of emotionally evoked theta rhythm in infancy: hedonic hypersynchrony. Electroencephalogr Clin Neurophysiol. 1971 Aug;31(2):157-65. doi: 10.1016/0013-4694(71)90186-6. No abstract available. PMID 4104705
- [Background] Vadiakas G, Oulis C, Berdouses E. Profile of non-nutritive sucking habits in relation to nursing behavior in pre-school children. J Clin Pediatr Dent. 1998 Winter;22(2):133-6. PMID 9643187
- See also: Excessive pressure to stop the NNS habits in children before 4 years of age can do more harm than good. — http://www.ada.org/~/media/ADA/Publications/Files/patient_77.pdf?la=en
- See also: British Orthodontic Society recommendations: dummy habits tend to stop before the adult teeth appear at age 6. Beyond 7-year age, problems with the teeth position may occur. — https://www.bos.org.uk/Public-Patients/Patient-Information-Leaflets
- See also: Paola Rosati - Poster on the proprioceptive benefits from NNS habits in children presented at the 1st Society for Interdisciplinary Placebo Studies (SIPS) conference, April 2-4, 2017, Leiden, Netherlands (abstract book N. 2.34 page 111) — http://docplayer.net/50505590-Program-abstract-book.html